CLINICAL TRIAL: NCT01441648
Title: Influence of Cosmetic Color Tinted Contact Lenses on the Ocular Surface
Status: Completed | Type: Observational
Sponsor: Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation (Other)
Collaborators: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 00-IRB-007-XD; Shen EP (Other: Buddhist Tzu Chi General Hospital, Taipei)
Record Dates: First submitted 2011-09-26; First posted 2011-09-28 (Estimated); Last update posted 2014-01-20 (Estimated); Status verified 2011-12

CONDITIONS: Conjunctival Infections, Irritations and Inflammations; Hypertrophy; Conjunctiva; Corneal Pannus; Corneal Epithelial Wound
Keywords: conjunctival injection; conjunctival papillary hypertrophy; pannus formation; corneal epitheliopathy; Schirmer test; Impression cytology; confocal microscopy; Scanning electronmicroscopy (SEM); bacterial adhesion determination
MeSH Terms: conditions — Inflammation; Hypertrophy | interventions — Contact Lenses, Extended-Wear

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- experimental group: (1) age 20-35 years old (2) myopia less than -6.00D and astigmatism less than -1.50D (3) previous soft contact lens wear discontinued for at least 2 weeks. Exclusion criteria includes: (1) subjects with previous Rigid Gas Permeable (RGP) wear (2) any ocular inflammation or infection, dry eye syndrome, glaucoma, ocular trauma or surgery, and topical medication instillation (3) diabetic mellitus (4) pregnancy (5) any corneal disorders or dystrophies.
  Interventions: Other: contact lens wear

INTERVENTIONS:
Other: contact lens wear — tinted contact lens wear
  Other Names: cosmetic colored contact lenses; Ciba Vision Freshlook

SUMMARY:
More than 1 million people worldwide wear soft contact lenses for refractive error correction. However, severe sight threatening complications due to contact lens wear such as contact lens-related microbial keratitis (CLMK) are about 1 per 2500 persons per year. The rate of infection increases drastically to 1 per 500 person per year if lenses were worn overnight. Recently, color tinted cosmetic soft contact lenses, which are essentially soft contact lenses with a color tinted annular ring, are gaining increasing popularity especially among the younger and Asian population desiring a change in iris color or the doll-eyed look. However, studies on the effect of these lenses on the ocular surface have been scarce. Recently, a report of 12 cases of lens-related microbial keratitis due to wear of the color tinted lenses have been reported. Others reported of decreased contrast sensitivity, increased higher order aberrations, and temporary changes in corneal topography due to color tinted lens wear. Nevertheless, comprehensive and prospective study has not yet been done. Thus, the purpose of this study is to conduct a prospective observational study to determine the influence of color tinted cosmetic contact lens wear both on visual performance and ocular surface alterations.

DETAILED DESCRIPTION:
3. Methods All subjects are required to fill out basic information and take a survey questionnaire before and after contact lens wear. Subjects will be examined and tested before being fitted to color tinted contact lens with slit-lamp biomicroscopy and fluorescein staining (Heig Strait, Germany), intraocular pressure measurement by pneumotonometery (Topcon® CT-80), refractometer (Topcon® KR-8900), uncorrected and best corrected Snellen visual acuity (UCVA and BCVA), Schirmir test 1, tear film break-up time (TBUT), corneal topography (Bausch & Lomb® Orb IIz), and endothelial cell density measurement by specular microscopy (Konan Noncon Robo-Sp-9000, USA). Exams are also performed at 1 week, 1, 3, and 6 months of lens wear. A special chart for all subjects is filled out during each visit During each exam, subjects will be observed for signs of conjunctival injection, conjunctival papillary hypertrophy, pannus formation, and corneal epitheliopathy. These signs are graded as shown in the table below.

Signs 0=Normal 1=Mild 2=Moderate 3=Severe Conjunctival Injection None Minimal Obvious Diffuse Papillae Size None <0.25mm 0.25-0.5mm >0.5mm Superficial Pannus No pannus 1 quadrant 2 quadrants >=3 quadrants Punctate Epitheliopathy None <1/3 of cornea 1/3-1/2 of cornea Confluent or with epithelial defect

Schirmir test 1 (basal secretion test) is performed for 5 minutes and considered abnormal if the filter strip wets <5 mm in length. TBUT of less than 10 seconds is considered abnormal.

Impression cytology will be performed before lens wear and at 3 and 6 months post lens wear at National Taiwan University. Nitrocellulose filter paper with the pore size of 0.22 μm (Millipore GSWP 04700, Billerica, MA, U.S.A.) are cut into strips (about 4x8 mm). After a drop of topical anesthetic (proparacaine 0.5 %) application, excess tears are gently absorbed by sterile cotton swabs. Nitrocellulose strip are placed on the surface of limbal conjunctiva. After applying light pressure, the paper strips are peeled off and immediately fixed in 95% alcohol. The strips are then stained using periodic acid-Schiff (PAS ; Sigma 395132, Hattiesburg, MS, USA) and examined under light microscopy at 40X magnification and graded by mask observers following Saini et al's criteria21 as follows. Grade 1: Small round epithelial cells with a nucleus to cytoplasm ration of 1:2. Large number of deeply positive cells present. A good confluent sheet of cells is usually obtained. Grade2: A good cell sheet consisting of larger polygonal epithelial cells with a decreased nucleocytoplasmic ration of 1:3. Goblet cells reduced in number, but still deeply PAS-positive. Grade 3: Larger polygonal cells with a further decrease in nucleus to cytoplasm ratio. Reduced number of goblet cells, with reduced staining. Grade 4: Larger polygonal basophilic cells with pyknotic nuclei. Intracellular keratin often demonstrable. Absent goblet cells. Only a few loose clumps were obtainable. Goblet cell density is also graded by counting the average number of cells per 100 epithelial cells in at least four high power fields (HPF). Grade 1: >30 goblet cells/ 4 HPF. Grade 2: 15-30 goblet cells/ 4 HPF. Grade 3: 5-15 goblet cells/ 4 HPF. Grade 4: <5 goblet cells/ 4 HPF.

In vivo confocal microscopy imaging of the cornea will be performed before lens wear and at 3 and 6 months post lens wear by one masked examiner on all subjects at National Taiwan University. One drop of 0.5% proparacaine solution and artificial tears was instilled immediately before each exam. After asking the patients to look straight ahead, an in vivo confocal microscope (Confoscan 3.4.1; Nidek Technologies, Padova, Italy) equipped with a standard 40x water-immersion front lens captured images of the full thickness of the central cornea automatically. Each examination took approximately 1 to 3 minutes and recorded 350 images at a distance of 1.5 and 4 μm on the z-axis between successive images. During each visit, measurements were repeated with 4 um z-interval for 3 times followed by 1.5 um z-interval for 3 times. Analysis of epithelial cells morphology, epithelial thickness, and stromal reaction follows that has been published by Chen et al22-24. Corneal nerve morphology and density will also be recorded and analyzed.

Used contact lenses will be place in the provided storage cases and brought back to check for completeness of lens with no tear or chipped pieces. The lenses are then used for further material analysis by scanning electromicroscopy (SEM) and bacterial adhesion determination with personal funding. For SEM, used lenses were fixed in half strength Karnovskys fixative ( 2% paraformaldehyde and 2.5% glutaraldehyde) after gentle washing. The fixative was removed and distilled water was added for rinsing. Rapid freezing with liquid nitrogen immersion was done before being placed under vacuum overnight. The concave side of samples was mounted on aluminum stubs and sputter-coated with gold for examination under SEM (JEOL Ltd, JSM 5300, Japan) at 15kV under various magnification. For bacterial adhesion determination, used lenses are collected in sterile plates and gently dipped three times in PBS before placement in eppendorf tubes containing 1ml PBS. The lenses are then macerated and serial dilutions up to 105 are done before plating onto Muller-Hinton agar. The agar plates are incubated overnight and colony forming units are counted the next day. Number of colonies multiplied by dilution factor divided by the volume plated will give the CFU/ml/per contact lens.

All data will be entered into Excel spreadsheet (Microsoft, Inc) and analyzed using SPSS software for Windows (11.0, SPSS, Inc.). Paired t-tests will be used to compare all parameters before and after wear of the color tinted contact lenses.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-35 years old
* myopia less than -6.00 D, Astigmatism less than 1.50 D
* previous soft contact lens wear discontinued for at least 2 weeks

Exclusion Criteria:

* subjects with previous Rigid Gas Permeable wear
* Any ocular surgery or topical medication
* dry eye syndrome
* glaucoma
* ocular trauma
* pregnancy
* any corneal disorders or dystrophies

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 1) age 20-35 years old (2) myopia less than -6.00D and astigmatism less than -1.50D (3) previous soft contact lens wear discontinued for at least 2 weeks. Exclusion criteria includes: (1) subjects with previous Rigid Gas Permeable wear (2) any ocular inflammation or infection, dry eye syndrome, glaucoma, ocular trauma or surgery, and topical medication instillation (3) diabetic mellitus (4) pregnancy (5) any corneal disorders or dystrophies.
Sampling Method: Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2011-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Comfort | during 6 month weart

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth P Shen, Principal Investigator — Buddhist Tzu Chi General Hospital, Taipei Branch
Locations (1):
- Buddhist Tzu Chi General Hospital, Taipei, New Taipei City, Taiwan